CLINICAL TRIAL: NCT02403180
Title: Comparative Assessment of Visual Performance Between DAILIES® AquaComfort Plus® (DACP) Multifocal (MF) and PROCLEAR 1 Day Multifocal (PROCLEAR 1D MF)
Brief Title: DAILIES® AquaComfort Plus® Multifocal (MF) - Comparative Assessment of Visual Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLW681-P001
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Results first posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Presbyopia
Keywords: Visual Performance
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DACP MF, then PROCLEAR 1D MF (Other): DACP MF (nelfilcon A) multifocal contact lenses worn in Period 1, followed by PROCLEAR 1D MF (omafilcon A) multifocal contact lenses worn in Period 2. Both products were worn bilaterally (in both eyes) for 5 ±1 days in a daily wear, daily disposable modality.
  Interventions: Device: DACP MF; Device: PROCLEAR 1D MF
- PROCLEAR 1D MF, then DACP MF (Other): PROCLEAR 1D MF (omafilcon A) multifocal contact lenses worn in Period 1, followed by DACP MF (nelfilcon A) multifocal contact lenses worn in Period 2. Both products were worn bilaterally (in both eyes) for 5 ±1 days in a daily wear, daily disposable modality.
  Interventions: Device: DACP MF; Device: PROCLEAR 1D MF

INTERVENTIONS:
Device: DACP MF — Nelfilcon A multifocal contact lenses
  Other Names: DAILIES® AquaComfort Plus® Multifocal (DACP MF); Nelfilcon A
Device: PROCLEAR 1D MF — Omafilcon A multifocal contact lenses
  Other Names: PROCLEAR® 1 DAY MULTIFOCAL (PROCLEAR 1D MF); Omafilcon A

SUMMARY:
The purpose of this study is to evaluate the visual performance of DACP MF and PROCLEAR 1D MF daily disposable contact lenses in an established presbyopic population.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent;
* Adapted soft contact lens wearer;
* Vision correctable to 20/30 [(0.2 logMAR (logarithm of the minimum angle of resolution)] or better in each eye at distance;
* Willing to wear lenses every day or for at least 5 days per week, 6 hours per day;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Currently wearing multifocal contact lenses;
* Currently wearing monovision;
* Ocular anterior segment infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear;
* Use of systemic or ocular medications which could contraindicate contact lens wear;
* Eye injury or surgery within 12 weeks prior to enrollment;
* Prior refractive surgery;
* Monocular (only 1 eye with functional vision) or fit with only 1 lens;
* Other protocol-specified exclusion criteria may apply.

Ages: 41 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, Study Director — Alcon, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one investigational center located in Spain.
Pre-assignment Details: This reporting group includes all enrolled participants (70).
Groups:
- DACP MF, Then PROCLEAR 1D MF: Nelfilcon A contact lenses were worn in Period 1, followed by omafilcon A contact lenses in Period 2. Both products were worn bilaterally (in both eyes) for 5 ±1 days in a daily wear, daily disposable modality.
- PROCLEAR 1D MF, Then DACP MF: Omafilcon A contact lenses were worn in Period 1, followed by nelfilcon A contact lenses in Period 2. Both products were worn bilaterally (in both eyes) for 5 ±1 days in a daily wear, daily disposable modality.
Period: Pre-Treatment Period
Arm/Group | DACP MF, Then PROCLEAR 1D MF | PROCLEAR 1D MF, Then DACP MF
Started | 36 | 34
Completed | 36 | 33
Not Completed | 0 | 1
Not completed — Withdrawal by subject prior to treatment | 0 | 1
Period: Period 1 (5 Days)
Arm/Group | DACP MF, Then PROCLEAR 1D MF | PROCLEAR 1D MF, Then DACP MF
Started | 36 | 33
Randomized | 36 | 33
Completed | 36 | 33
Not Completed | 0 | 0
Period: Period 2 (5 Days)
Arm/Group | DACP MF, Then PROCLEAR 1D MF | PROCLEAR 1D MF, Then DACP MF
Started | 36 | 33
Completed | 36 | 32
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention to treat, defined as the set of all randomized participants.
Groups:
- DACP MF, Then PROCLEAR 1D MF: Nelfilcon A contact lenses were worn in Period 1, followed by omafilcon A contact lenses in Period 2.
- PROCLEAR 1D MF, Then DACP MF: Omafilcon A contact lenses were worn in Period 1, followed by nelfilcon A contact lenses in Period 2.
- Total: Total of all reporting groups
Arm/Group | DACP MF, Then PROCLEAR 1D MF | PROCLEAR 1D MF, Then DACP MF | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (4.67) | 50.4 (3.88) | 51.1 (4.32)
Age, Customized [Number; unit: participants]
  41-50 years | 15 | 20 | 35
  51-60 years | 20 | 13 | 33
  61-65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 48
  Male | 14 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Stereoacuity at Near After 5+/-1 Days of Contact Lens Wear
Description: Stereoacuity (SA) is the ability to detect differences in distance (depth perception). Near SA was measured at a distance of 40 cm using the Howard-Dolman system. A lower SA value indicates better depth perception.
Time Frame: Day 5, each product
Population: Intention to treat participants with non-missing observations
Measure: Mean (Standard Deviation); unit: arcsec
Groups:
- Proclear 1 Day MF: Omafilcon A contact lenses were worn for 5 days in Period 1 or Period 2.
- DACP MF: Nelfilcon A contact lenses were worn for 5 days in Period 1 or Period 2.
Arm/Group | Proclear 1 Day MF | DACP MF
Number analyzed (Participants) | 69 | 68
arcsec | 40.6 (11.67) | 30.7 (8.67)

2. Secondary Outcome: Mean Area of Focus Under the Mean Defocus Curve After 5 +/- 1 Days of Contact Lens Wear
Description: Visual acuity was measured with contact lenses in place using an Early Treatment Diabetic Retinopathy Study (ETDRS) high contrast logMAR chart under well-lit conditions. Trial Lenses of different spherical powers (+2.00 diopter to -5.00 diopter) were placed in front of the eyes to produce varying levels of defocus, and logMAR acuity at each defocus value was recorded. The area under the defocus curve (AUC) was calculated via the trapezoidal rule for the entire study population by treatment using a 0.3 logMAR threshold for intermediate from -2.00 D (50cm) to -0.50 D (2m) and near from -4.00 D (25cm) to -2.00 D (50cm). A higher value indicates a bigger area of focus.
Time Frame: Day 5, each product
Population: Intention to treat participants with non-missing observations
Measure: Mean (Standard Deviation); unit: diopter*logMar
Arm/Group | Proclear 1 Day MF | DACP MF
Number analyzed (Participants) | 69 | 68
diopter*logMar
  for the Near Region | 0.04 (0.051) | 0.07 (0.061)
  for the Intermediate Region | 0.17 (0.092) | 0.21 (0.077)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study from the time of first lens fitting, throughout 10 days (+/- 2 days) of lens wear.
Description: AEs were defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs, whether or not related to the medical device, obtained through solicited and spontaneous comments from all exposed participants and reported based on the treatment received. Ocular AEs are presented for both eyes combined.
Arm/Group | Proclear 1 Day MF | DACP MF
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/69
Other Adverse Events (participants affected / at risk) | 0/69 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.